CLINICAL TRIAL: NCT03157011
Title: Evaluation of the Prevalence of Functional Digestive Disorders During Primary Sjögren Gougerot Syndrome
Acronym: GASTRO-SGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: I16033 (GASTRO-SGS)
Record Dates: First submitted 2017-05-02; First posted 2017-05-17 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-07

CONDITIONS: Sjogren's Syndrome; Digestive System Abnormalities
Keywords: Primary Sjögren syndrome - Digestive symptoms
MeSH Terms: conditions — Sjogren's Syndrome; Digestive System Abnormalities

STUDY DESIGN:
Intervention Model Description: Global symptom score (GSS) questionary . This questionnaire has the advantage of grading the severity of These digestive symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Global symptom score (GSS) questionary (Experimental): systematic research of digestive symptoms in patients with SGSp with Global symptom score (GSS) questionary.
  Interventions: Other: Global symptom score (GSS) questionary

INTERVENTIONS:
Other: Global symptom score (GSS) questionary — systematic research of digestive symptoms in patients with SGSp with Global symptom score (GSS) questionary, which allowed to grades severity of 10 digestive symptoms (absent, mild, moderate, or severe), asthenia and fever.

SUMMARY:
the investigators propose to carry out a prospective study consisting of a systematic research of digestive symptoms in patients with SGSp with the validated Global symptom score (GSS) questionnaire, which allowed to grades severity of 10 digestive symptoms (absent, mild, moderate, or severe), asthenia and fever.

DETAILED DESCRIPTION:
Primary Sjögren syndrome (SGSp) is an autoimmune disease defined by the association of sicca syndrome in the absence of other connective tissues (ie rheumatoid arthritis, systemic lupus erythematosus, scleroderma, dermatopolymyositis). SGSp is complicated by several visceral involvements (pulmonary, renal, neurological, systemic vasculitis ...) and by a chronic alteration of the quality of life related to asthenia, chronic pain and sicca syndrome. Two European-validated scales are currently used in daily clinical practice to assess these two facets of the disease, respectively EUSSAR Sjogren's Syndrome Patient Reported Index (ESSPRI) and ESSDAI (EULAR Sjögren's Syndrome Disease Activity Index). Neither of these two scores evaluate the digestive impairment. Indeed, digestive complaints have been evaluated in a few studies, with a prevalence of 30 to 65%. The precise etiopathogeny of such digestive involvements remains unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SGSp according to revised American-European criteria
* Patients 18 years of age or older
* Patients affiliated to the French social security care system.

Exclusion Criteria:

* Patients under measure of maintenance of justice.
* Patients unable to understand or to participate to the study.
* Child and major patients making the object of a measure of lawful protection.
* Patients deprived of freedom.
* Concomitant interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of functional digestive symptoms during SGSp | 19 months (End of study)
  Measure the prevalence of functional digestive symptoms during SGSp globally and as a function of the duration of the disease

SECONDARY OUTCOMES:
Prevalence of each GSS symptom | 19 months (End of study)
  Measure the prevalence of each GSS symptom and its severity during the pSGS, globally and depending on the duration of disease
Prevalence of stomach digestive symptoms | 19 months (End of study)
  Measure the prevalence of each GSS symptom and its severity during the pSGS, globally and depending on the duration of disease
Association between the presence of digestive disorders and SGSp activity | 19 months (End of study)
  Determine the possible association between the presence of digestive disorders (each symptom) and SGSp activity, painfulness experienced by the patient, anti-SSA antibody, and / or SSB
Association between the presence of digestive symptoms, the existence of a sicca syndrome at the time of screening | 19 months (End of study)
  Determine the possible association between the presence of digestive symptoms, the existence of a sicca syndrome at the time of screening, neurological involvement, pulmonary involvement, parotiditis, depressive disorders, fibromyalgia, hypergammaglobulinemia
Digestive disorders | 19 months (End of study)
  Describe the digestive disorders discovered by the digestive explorations generated by the existence of digestive symptoms, in accordance with the usual rules of good practice

CONTACTS AND LOCATIONS:
Overall Officials: ANNE-LAURE FAUCHAIS, PH, Principal Investigator — University Hospital, Limoges
Locations (1):
- University Hospital, Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parreau S, Jacques J, Dumonteil S, Palat S, Geyl S, Gondran G, Bezanahary H, Liozon E, Azais J, Colombie S, Jauberteau MO, Loustaud-Ratti V, Ly KH, Fauchais AL. Abdominal symptoms during Sjogren's syndrome: a pilot study. Adv Rheumatol. 2021 Jan 19;61(1):5. doi: 10.1186/s42358-021-00164-w. PMID 33468262